CLINICAL TRIAL: NCT00487851
Title: Endoscopic Strategy Versus Surgical by Pass in Nonresectable Periampullary Cancer
Brief Title: Comparing Endoscopic Based Stent Strategy Versus Bypass Surgery in Non-resectable Periampullary Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Farshad Frozanpor, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006/2:3
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Pancreatic Neoplasms; Biliary Tract Neoplasms; Duodenal Neoplasms
Keywords: Pancreatic; cancer; Periampullay; Neoplasms; Biliary; Duodenal; Jaundice; obstruction; pancreas cancer; Pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms; Duodenal Neoplasms; Neoplasms; Jaundice; Bites and Stings | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Endoscopic treatment strategy
  Interventions: Procedure: endoscopic strategy
- 2 (Active Comparator): Surgical treatment strategy
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — hepaticojejunostomy and gastroenterostomy
  Arms: 2
Procedure: endoscopic strategy — Stent insertion
  Arms: 1

SUMMARY:
Randomized study comparing endoscopic stent insertion strategy versus double-bypass surgery in non-resectable periampullary cancer

DETAILED DESCRIPTION:
Experience shows that patients with advanced periampullary cancer suffer not only from jaundice but in 25 -30% of cases also duodenal stricture with nausea, vomiting and nutritional difficulties. Ten years ago, the only palliative treatment for these patients was a bypass operation for bile flow and intestinal passage. This operation was often associated with a high morbidity. Developments in endoscopic treatments allow palliation with lower morbidity. However, stent treatment is not free of problems like stent dysfunction. During the last ten years, anesthesia and surgical techniques have developed which allow lower postoperative morbidity compared to earlier treatments. A total of 70 patients were randomized to surgery with hepaticojejunostomy on Roux loop and gastrojejunostomy or endoscopic treatment with self-expanding metallic stent in the bile duct and so-called duodenal stent. Based on the inclusion of 70 patients, we expected a 20% difference in some of the primary variables with a power of 80%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a locally advanced periampullary neoplastic process with extrahepatic bile duct obstruction.
* The patient tumor burden and general condition should be such that treatment related morbidity and mortality is calculated as "reasonable" and both treatment strategies are considered "applicable".

Exclusion Criteria:

* Non consent.
* The patients' general condition will not tolerate either treatment (strategy).
* Previous laparotomy or laparoscopy.
* Life expectancy < 3 months.
* Inability to participate (language, social, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Primary outcome consist of a composite score (i.e. number of hospitalizations, episodes of cholangitis, degree of jaundice, other complications requiring therapeutic interventions). Secondary outcome are QoL,hospital stay and health economic burden. | 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Farshad Frozanpor, Principal Investigator — Karolinska institut Huddinge
Locations (1):
- Karolinksa university hospital, Huddinge, Sweden